CLINICAL TRIAL: NCT03571295
Title: A Comparison of Direct Laryngoscopy and King Vision® aBlade™ Videolaryngoscopy in Paediatric Airway Management: Success Rate and Learning Curve of Trainee Anaesthetists
Brief Title: Comparison of Videolaryngoscopy and Direct Laryngoscopy in Pediatric Airway Management
Acronym: LearnaBlade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Consultant, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Learn a Blade 1.0
Record Dates: First submitted 2018-05-22; First posted 2018-06-27 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Airway Management; Videolaryngoscopy
Keywords: pediatric airway management; learning curve

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- videolaryngoscopy (Experimental)
  Interventions: Device: King Vision aBlade
- direct laryngoscopy (Experimental)
  Interventions: Device: direct laryngoscopy

INTERVENTIONS:
Device: King Vision aBlade — endotracheal intubation performed with King Vision aBlade
  Arms: videolaryngoscopy
Device: direct laryngoscopy — endotracheal intubation performed with direct laryngoscopy
  Arms: direct laryngoscopy

SUMMARY:
The investigators intended to evaluate first success rate and learning curve of trainee anesthetists performing direct and videolaryngoscopy in pediatric airway management.

DETAILED DESCRIPTION:
After obtaining written informed consent of 10 trainee anesthetists with non less than 24 months and not exceeding 60 months residency, use of the King Vision aBlade videolaryngoscope was demonstrated by presenting a 2 min instruction video. First endotracheal intubation by each trainee anesthetist was randomly allocated to either direct (DL) or King Vision aBlade videolaryngoscopy (KingVL). Then order of laryngoscopy type was alternating at least each trainee anesthetists performed 10 DL and 10 KingVL endotracheal intubations.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to 2
* written informed consent from both legal guardians
* children who were scheduled for nonemergency surgery with requirement of endotracheal intubation

Exclusion Criteria:

* known or predicted difficult airway
* increased risk for pulmonary aspiration

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
first attempt success rate of endotracheal intubation | operation day
  yes/no

SECONDARY OUTCOMES:
total time for successful intubation | operation day
  in sec

OTHER OUTCOMES:
failure category of the first attempt | operation day
  First attempt failed when esophageal intubation or oxygen desaturation < 90% occurred.

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg - Universität, Mainz, Rhineland-Palatinate, Germany